CLINICAL TRIAL: NCT05777915
Title: Preliminary Studies to the SOSteniamoci Project: Usability Study
Brief Title: SOSteniamoci: Usability Study
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 03C211
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Internet-based Intervention
MeSH Terms: interventions — User-Centered Design

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Usability testing — Usability testing

SUMMARY:
The goal of this observational study is to test the usability of the SOSteniamoci platform, culturally adapted from the Lithuanian context, for informal caregivers in Italy.

The main goals were to (1) collect qualitative and quantitative data on usability and (2) identify usability problems. A balanced gender-age sample of 10 individuals meeting the inclusion criteria was consecutively recruited online. The think-aloud testing method, the system usability scale, and an ad hoc semi-structured interview were employed to determine the overall system usability.

DETAILED DESCRIPTION:
The study employed a mixed methods sequential explanatory design approach, comprising the following end-user testing: (1) a phase of collection and analysis of measures of performance employing the think-aloud method, (2) a phase of collection and analysis of quantitative data through the use of a System Usability Scale (SUS) and (3) a phase of collection and analysis of qualitative data through the use of an ad hoc semi-structured interview to further explain the results obtained in the earlier stages.

Ten individuals who showed interest in participating in the SOSteniamoci project by writing to the email address behind the official website (https://www.iterapi.se/sites/sosteniamoci/) were consecutively asked to take part in the usability test based on the inclusion criteria. A balanced gender-age sampling was used to best reflects the heterogeneity of the population.

As a result of the COVID-19 pandemic, all procedures were performed online (completion time: 45 mins, on average). First, each participant received an email with a) the link to the online meeting, including the date and time, and b) the link and access credentials of the SOSteniamoci platform. Before starting the usability test, the researcher provided detailed information about the test procedures and described the purpose of the computer-based self-management system. Participants were then asked to give their online informed consent, provide demographic information, and report on their level of comfort with computers and the Internet.

They were also asked if they had already taken a usability test before. All participants were assigned a unique ID unrelated to their identity. Personal data were linked only to this unique ID and stored in a secure online platform accessible only by the research team and protected by a password.

ELIGIBILITY:
Inclusion criteria:

* age >18 years
* be able to read and speak the Italian language
* have basic computer skills and Internet access
* own a computer or a compatible device
* having provided informed consent to participate.

Exclusion criteria:

- presentation of self-reported visual, hearing, or cognitive impairments preventing the participant from following the instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Informal caregivers of a person with a chronic disease
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Score of System Usability Scale (SUS) | baseline
  10-item scale with final score between 0 and 100

CONTACTS AND LOCATIONS:
Overall Officials: Giada Pietrabissa, PhD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
There is not plan to make IPD available.